CLINICAL TRIAL: NCT06444282
Title: Optimization and Implementation Trial of a User-Centered Emergency Care Action Plan for Infants with Medical Complexity
Brief Title: Emergency Care Action Plans for Infants with Medical Complexity
Acronym: ECAP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Christian Pulcini, Principal Investigator, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1K23HD109469-01 (NIH); K23HD109469-01 (NIH)
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Children with Medical Complexity; Child, Only; Infant Morbidity; Infant Conditions; Utilization, Health Care; Emergencies; Chronic Condition
MeSH Terms: conditions — Patient Acceptance of Health Care; Emergencies; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emergency Care Action Plan (Experimental): An Emergency Care Action Plan (ECAP) is a brief, pre-populated summary of suggested emergency management for children with medical complexity, embedded in the electronic health record.
  Interventions: Other: Emergency Care Action Plan
- Standard Care (No Intervention): The current standard of care does not include emergency care planning.

INTERVENTIONS:
Other: Emergency Care Action Plan — An Emergency Care Action Plan (ECAP) is a brief, pre-populated summary of suggested emergency management for children with medical complexity, embedded in a patient's electronic health record for access by providers in an emergency. Patients/families will have digital access to the ECAP and be given a paper copy. The patient's care team and caregiver(s) (parent/legal guardian) will collaborate to create an individualized ECAP containing the following content: caregiver contact information, patient summary, anticipated emergency presentations with suggested management, problem list (emergency relevant only), medication list, technology dependence, baseline important physical exam findings, baseline vital signs, allergies, advance directive information, contact information for established care providers, and other important information.
  Arms: Emergency Care Action Plan

SUMMARY:
An Emergency Care Action Plan (ECAP) is a tool intended to be helpful to providers when treating a child with complex medical needs during an emergency. Once created, ECAPs are added to the Electronic Health Record (EHR), shared with the child's caregiver(s), and kept up by all of those involved in a child's care.

The goal of this study is to measure important health outcomes (ex. inpatient days, emergency department visits) in terms of the use of the ECAP for infants discharged from the Neonatal Intensive Care Unit (NICU). This study will also measure other real-time potential challenges related to the use of the ECAP including, but not limited to, if it is being used, if providers and caregivers want to use it, and if they keep using it over a long period of time.

DETAILED DESCRIPTION:
National expert recommendations and human-centered design principles were used to optimize an Emergency Care Action Plan (ECAP) for infants with medical complexity. This study will implement and monitor the effectiveness and feasibility of the optimized Emergency Care Action Plan for infants with medical complexity. The primary objective is to determine the effectiveness of a user-centered Emergency Care Action Plan for infants with medical complexity on emergency health care utilization and cost metrics. The secondary objective is to monitor and evaluate barriers and facilitators to the current and widespread implementation of a user-centered Emergency Care Action Plan for infants with medical complexity.

Research participants will be assigned by chance to receive an ECAP or standard care. Caregivers (parent/legal guardian) of infant participants will be asked to complete periodic surveys during a one-year feasibility trial period. If assigned, caregivers will be asked to help with the process of creating an ECAP for their child.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 to 6 months
* Admitted to the University of Vermont Medical Center Neonatal Intensive Care Unit (NICU)
* Meets or is expected to meet Children with Medical Complexity status as determined by the treating NICU clinician and defined as "children with multiple significant chronic health problems including multiple organ systems, which result in functional limitations, high health care needs or utilization, and often require need for, or use of, medical technology."

Exclusion Criteria:

* Does not have a caregiver participant who agrees to their participation in the study to complete follow-up surveys
* Does not intend to use University of Vermont Health Network and affiliated sites for care during the one-year trial period

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2027-08-08 (Estimated); Study Completion 2028-08-08 (Estimated)

PRIMARY OUTCOMES:
Inpatient hospitalization | Day 0 (NICU discharge) to Month 12
  Number of inpatient hospital days

SECONDARY OUTCOMES:
Avoidance of ED visits | Day 0 (NICU discharge) to Month 12
  Caregiver's perceived avoidance of emergency department (ED) visits for their child
Number of ED visits | Day 0 (NICU discharge) to Month 12
  Number of emergency department (ED) visits
ED length of stay | Day 0 (NICU discharge) to Month 12
  Emergency department (ED) length of stay
Interfacility transfers | Day 0 (NICU discharge) to Month 12
  Number of interfacility transfers
Caregiver stress | Day 0 (NICU discharge) to Month 12, assessed at quarterly intervals (Month 3, 6, 9, 12)
  Caregiver perceived stress measured using the University of Washington Caregiver Stress Scale 3 item short form for caregivers of children with serious health conditions.
Caregiver self-efficacy | Day 0 (NICU discharge) to Month 12, assessed at quarterly intervals (Month 3, 6, 9, 12)
  Caregiver self-efficacy in health care information or decision making and symptoms identification or management measured using the Parent Measure of Self-Efficacy Managing a Child's Medication and Treatments, adapted from the Patient-Reported Outcomes Measurement Information Systems (PROMIS).

OTHER OUTCOMES:
Cost | Day 0 (NICU discharge)-Month 12
  Costs for healthcare services received
Implementation outcomes | Day 0 (NICU discharge) to Month 12, assessed at quarterly intervals (Month 3, 6, 9, 12)
  Caregiver and provider perspectives on acceptability, adoption, appropriateness, feasibility, useability, and sustainability of Emergency Care Action Plans prior to and throughout implementation will be accessed, in addition to barriers/facilitators to implementation and suggestions for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Christian D Pulcini, MD, MEd, MPH, Principal Investigator — University of Vermont Larner College of Medicine, University of Vermont Medical Center
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after de-identification will be shared (text, tables, figures and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 26 months following article publication.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research for individual participant data meta analysis. Proposals may be submitted up to 36 months following article publication. Proposals must be reviewed and approved by an independent review committee identified for this purpose. Proposals should be directed to Christian.Pulcini@uvmhealth.org.

REFERENCES:
- [Background] Pulcini CD, Rubin DM. Flipping the Script on Emergency Care for Children With Medical Complexity. Pediatrics. 2019 Sep;144(3):e20183905. doi: 10.1542/peds.2018-3905. No abstract available. PMID 31439622
- [Background] Pulcini CD, Dubuque A, Lamberson M, Macy ML, Mistry RD, Pruitt CM, Schnadower D, Zorc JJ, Stevens MW. Pediatric Emergency Medicine Physicians' Perspectives on Emergency Care of Children With Medical Complexity: A Multi-institution Mixed-Methods Assessment. Pediatr Emerg Care. 2022 Aug 1;38(8):e1423-e1427. doi: 10.1097/PEC.0000000000002712. Epub 2022 Apr 18. PMID 35436769
- [Background] Pulcini CD, Belardo Z, Ketterer T, Zorc JJ, Mollen CJ. Improving Emergency Care for Children With Medical Complexity: Parent and Physicians' Perspectives. Acad Pediatr. 2021 Apr;21(3):513-520. doi: 10.1016/j.acap.2020.09.006. Epub 2020 Sep 15. PMID 32947009
- [Background] Pulcini CD, Coller RJ, Houtrow AJ, Belardo Z, Zorc JJ. Preventing Emergency Department Visits for Children With Medical Complexity Through Ambulatory Care: A Systematic Review. Acad Pediatr. 2021 May-Jun;21(4):605-616. doi: 10.1016/j.acap.2021.01.006. Epub 2021 Jan 21. PMID 33486099
- [Background] Pulcini CD, Coller RJ, Macy ML, Alpern E, Harris D, Rodean J, Hall M, Chung PJ, Berry JG. Low-Resource Emergency Department Visits for Children With Complex Chronic Conditions. Pediatr Emerg Care. 2022 Feb 1;38(2):e856-e862. doi: 10.1097/PEC.0000000000002437. PMID 34009894
- [Derived] Palaza A, Callas P, Dayan PS, Kuo DZ, Riney L, Spencer SP, Stapleton R, Stevens M, Studts CR, Pulcini CD. Randomised hybrid type 1 pilot trial evaluating preliminary effectiveness and implementation of an emergency care action plan (ECAP) for infants with medical complexity within a rural health network: a study protocol. BMJ Open. 2025 Oct 6;15(10):e106842. doi: 10.1136/bmjopen-2025-106842. PMID 41057174